CLINICAL TRIAL: NCT03883243
Title: Monitoring and Telecoaching of Physical Activity in Patients With Stage III and IV Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Wim Janssens, Prof. Dr. Wim Janssens, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S62244
Record Dates: First submitted 2019-02-04; First posted 2019-03-20 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Exercise; Neoplasms
Keywords: Telecoaching; Physical activity; Lung cancer
MeSH Terms: conditions — Motor Activity; Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective non-randomised controlled pilot study. 16 patients will be included in the intervention group and 16 patients will be included in a matched control group receiving only usual care.
Masking Description: Patients are evenly divided into the telecoaching group or usual care group according to owning a smartphone and their affinity with it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will only receive a brochure explaining the importance of physical activity with recommendations to improve it.
- Telecoaching (Experimental): Patients will receive a brochure explaining the importance of physical activity with recommendations to improve it. Next to this patients will receive the telecoaching intervention in which a coaching application linked to a step counter is installed on the patients smartphone, which will weekly give a new physical activity goal to improve the amount of steps per day for 8 weeks.
  Interventions: Device: Telecoaching

INTERVENTIONS:
Device: Telecoaching — A telecoaching application linked to a step counter will be installed on a patients smartphone for 8 weeks. The application shows a daily goal (expressed as amount of steps per day) to the patient. This goal is weekly revised and patients themselves are able to increase the goal every week with 500 or 1000 steps/day. Every evening, they are able to check the daily feedback platform, which gives them insights in their physical activity pattern of the day and previous weeks. At a regular basis, 'tip of the day' messages appear as a pop-up, to keep patients motivated.
  Arms: Telecoaching

SUMMARY:
This study is a prospective non-randomised control study to evaluate the efficacy of a physical activity promotion program on the experience of physical activity in patients with stage III and IV non-small cell lung cancer (NSCLC) with documented disease control (stable disease, partial or complete response defined by RECIST V1.1) at least 6 months after start of first line treatment.

The trial will consist of 4 visits. An outpatient clinic visit in which the eligible patients are invited (V1), a screenings visit (V2), a third visit (V3) at which the patients will be divided into the intervention or the control group, according to owning a smartphone and their affinity with it, followed by the start of the intervention consisting of 8 weeks telecoaching by means of an application and step counter and a final visit (V4) 8 weeks after starting up the intervention.

DETAILED DESCRIPTION:
The objective of this pilot study is to investigate if physical activity can be improved by telecoaching in patients with advanced stages of lung cancer in remission. We hypothesize that a smartphone application, designed for a population with respiratory symptoms, will increase daily physical activity, which translates into significant improvements on quality of life. This uncontrolled pilot study will therefore address if a 8-week PA promotion telecoaching program in addition to usual care has the potential to improve physical activity and quality of life in patients with lung cancer for a limited burden and at low cost.

This trial consists of 4 visits:

Visit 1 (V1, outpatient clinic):

Patients will be screened for inclusion in the study during follow up visits in the outpatient lung cancer clinic. If oncological check-up 6 months after starting initial lung cancer treatment demonstrates objective response (partial response or complete response defined by RECIST V1.1) the patient is asked to join the study. If the patient wants to join the study a screening visit (V2) will be planned.

Visit 2 (V2, screening visit (run-in)):

During V2 all eligible patients who have signed the informed consent will enter the run in epoch of 1 to 2 weeks.

Patients are asked about their medical history (baseline demographic data) and their previous respiratory treatment including their oncological stage and type. Co-morbidities will also be assessed and a basic lung function will be performed.

On V2 patient will receive a Dynaport movemonitor to wear one week before V3. For patients where the run in period is more than one week, they will receive a telephone reminder to wear a PROactive monitor. Patients are instructed to wear the device during waking hours. A measurement of more than 8 hours of wearing time will be defined as a 'valid day). The tri-axial accelerometer will captured steps waked per day, movement intensity and time spent in sitting, lying walking and high-intense activities.

Visit 3 (V3, baseline, allocation):

Patients will complete the web-based version of the clinical visit of the PROactive questionnaire. Two six-minutes walk tests will be performed and the patient will complete 2 quality of life questionnaires (SGRQ and QLQ-C30). During V3, the patients are divided into either control (usual care) or telecoaching group based on personal preferences and the abilities of using and having a smartphone.

Patients in both groups will receive a brochure during this visit explaining the importance of physical activity with recommendations to improve it. This brochure will be discussed together with the patients.

In the intervention group patients will recieve the telecoaching intervention consisting of the following components: 1: motivational interview with the investigator discussing motivation, barriers, favourite activities and strategies to become more active; 2: a pedometer giving direct feedback on the amount of steps; 3: the coaching application linked to the pedometer, which will be installed on the patient's smartphone and which will be coaching the patient for 8 weeks by means of improving the amount of steps per day. 4: telephone contact when a patient is non-compliant with either the use of the coaching intervention or with achieving the physical activity goals for 2 consecutive weeks.

All patients will be equipped with the Dynaport movemonitor one week before V4 and will be instructed to wear the monitor for 7 consecutive days.

Visit 4 (V4, end of the study, 8 weeks post allocation):

V4 is the end of the study. All assessments performed on V3 will be repeated during this study visit.

ELIGIBILITY:
1. Patients diagnosed with stage III or stage IV NSCLC who have a documented disease control (stable disease, partial or complete response defined by RECIST V1.1) at least 6 months after start of first line treatment. Stage III patients can only be included, if first line treatment consisted of concurrent chemoradiotherapy and a consolidation immunotherapy if indicated (if PDL1 > 1% and no potential contraindications for immunotherapy). Stage IV patients, should have received only immunotherapy (PDL1 > 50%) or a treatment of at least 4 cycles of a platinum based chemotherapy with or without immunotherapy. Maintenance therapy with chemotherapy and/or immunotherapy and administration of local radiotherpy is allowed. Patients with objective response can be included in the study until 2 years after starting up initial treatment.
2. > 18 years
3. Patients who are able to engage in a remote coaching program through the use of a smartphone

Exclusion criteria:

1. Patients actively participating in a pulmonary rehabilitation program
2. Patients with sequential chemoradiotherapy for stadium III non-small cell lung cancer
3. The presence of orthopedic problems not allowing an increase in PA levels

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in average daily number of steps | 8 weeks
  To assess the impact of a telecoaching program on physical activity in patients with stage III and IV NSCLC in addition to usual care. This will be measured by the Dynaport movemonitor (Dynaport®), as the change in average daily number of steps at baseline (1 week preceding V3) and at the end (1 week preceding V4) in the intervention and the control group.

SECONDARY OUTCOMES:
Change in health status | 8 weeks
  Change in health status assessed by QLQ-C30 (Cancer quality of life questionnaire) at baseline (1 week preceding) and at the end (1 week preceding) in the intervention and the control group.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level
Change in exercise capacity | 8 weeks
  Change in exercise capacity by 6 minutes walking distance at baseline and at the end in the intervention and the control group.

OTHER OUTCOMES:
Pro Active questionnaire | 8 weeks
  symptoms and difficulties perceived during exercise: Absolute difference in points from baseline values
health related quality of life: SGRQ | 8 weeks
  measured by SGRQ: proportion of patients with a minimal change of -4 points on SGRQ

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, Prof. Dr., Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
No, because this is a pilot trail we are not going to share the data with other researchers.

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Zappa C, Mousa SA. Non-small cell lung cancer: current treatment and future advances. Transl Lung Cancer Res. 2016 Jun;5(3):288-300. doi: 10.21037/tlcr.2016.06.07. PMID 27413711
- [Background] Dela Cruz CS, Tanoue LT, Matthay RA. Lung cancer: epidemiology, etiology, and prevention. Clin Chest Med. 2011 Dec;32(4):605-44. doi: 10.1016/j.ccm.2011.09.001. PMID 22054876
- [Background] Johnsen AT, Petersen MA, Pedersen L, Groenvold M. Symptoms and problems in a nationally representative sample of advanced cancer patients. Palliat Med. 2009 Sep;23(6):491-501. doi: 10.1177/0269216309105400. Epub 2009 May 14. PMID 19443525
- [Background] Thompson E, Sola I, Subirana M. Non-invasive interventions for improving well-being and quality of life in patients with lung cancer--a systematic review of the evidence. Lung Cancer. 2005 Nov;50(2):163-76. doi: 10.1016/j.lungcan.2005.06.004. Epub 2005 Aug 31. PMID 16137786
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Kraus WE, Bittner V, Appel L, Blair SN, Church T, Despres JP, Franklin BA, Miller TD, Pate RR, Taylor-Piliae RE, Vafiadis DK, Whitsel L; American Heart Association Physical Activity Committee of the Council on Lifestyle and Metabolic Health, Council on Clinical Cardiology, Council on Hypertension, and Council on Cardiovascular and Stroke Nursing. The National Physical Activity Plan: a call to action from the American Heart Association: a science advisory from the American Heart Association. Circulation. 2015 May 26;131(21):1932-40. doi: 10.1161/CIR.0000000000000203. Epub 2015 Apr 27. No abstract available. PMID 25918126
- [Background] Fong DY, Ho JW, Hui BP, Lee AM, Macfarlane DJ, Leung SS, Cerin E, Chan WY, Leung IP, Lam SH, Taylor AJ, Cheng KK. Physical activity for cancer survivors: meta-analysis of randomised controlled trials. BMJ. 2012 Jan 30;344:e70. doi: 10.1136/bmj.e70. PMID 22294757
- [Background] Lee IM. Physical activity and cancer prevention--data from epidemiologic studies. Med Sci Sports Exerc. 2003 Nov;35(11):1823-7. doi: 10.1249/01.MSS.0000093620.27893.23. PMID 14600545
- [Background] Granger CL, Connolly B, Denehy L, Hart N, Antippa P, Lin KY, Parry SM. Understanding factors influencing physical activity and exercise in lung cancer: a systematic review. Support Care Cancer. 2017 Mar;25(3):983-999. doi: 10.1007/s00520-016-3484-8. Epub 2016 Nov 29. PMID 27900549
- [Background] Michaels C. The importance of exercise in lung cancer treatment. Transl Lung Cancer Res. 2016 Jun;5(3):235-8. doi: 10.21037/tlcr.2016.03.02. PMID 27413700
- [Background] Kuehr L, Wiskemann J, Abel U, Ulrich CM, Hummler S, Thomas M. Exercise in patients with non-small cell lung cancer. Med Sci Sports Exerc. 2014 Apr;46(4):656-63. doi: 10.1249/MSS.0000000000000158. PMID 24042307
- [Background] Cramp F, Byron-Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD006145. doi: 10.1002/14651858.CD006145.pub3. PMID 23152233
- [Background] Bade BC, Thomas DD, Scott JB, Silvestri GA. Increasing physical activity and exercise in lung cancer: reviewing safety, benefits, and application. J Thorac Oncol. 2015 Jun;10(6):861-71. doi: 10.1097/JTO.0000000000000536. PMID 25831230
- [Background] Conn VS, Hafdahl AR, Brown SA, Brown LM. Meta-analysis of patient education interventions to increase physical activity among chronically ill adults. Patient Educ Couns. 2008 Feb;70(2):157-72. doi: 10.1016/j.pec.2007.10.004. Epub 2007 Nov 26. PMID 18023128
- [Background] Glynn LG, Hayes PS, Casey M, Glynn F, Alvarez-Iglesias A, Newell J, OLaighin G, Heaney D, O'Donnell M, Murphy AW. Effectiveness of a smartphone application to promote physical activity in primary care: the SMART MOVE randomised controlled trial. Br J Gen Pract. 2014 Jul;64(624):e384-91. doi: 10.3399/bjgp14X680461. PMID 24982490
- [Background] Institute of Medicine (US) Committee on Evaluating Clinical Applications of Telemedicine; Field MJ, editor. Telemedicine: A Guide to Assessing Telecommunications in Health Care. Washington (DC): National Academies Press (US); 1996. Available from http://www.ncbi.nlm.nih.gov/books/NBK45448/ PMID 20845554
- [Background] Cox A, Lucas G, Marcu A, Piano M, Grosvenor W, Mold F, Maguire R, Ream E. Cancer Survivors' Experience With Telehealth: A Systematic Review and Thematic Synthesis. J Med Internet Res. 2017 Jan 9;19(1):e11. doi: 10.2196/jmir.6575. PMID 28069561
- [Background] McCue M, Fairman A, Pramuka M. Enhancing quality of life through telerehabilitation. Phys Med Rehabil Clin N Am. 2010 Feb;21(1):195-205. doi: 10.1016/j.pmr.2009.07.005. PMID 19951786
- [Background] Grustam AS, Severens JL, De Massari D, Buyukkaramikli N, Koymans R, Vrijhoef HJM. Cost-Effectiveness Analysis in Telehealth: A Comparison between Home Telemonitoring, Nurse Telephone Support, and Usual Care in Chronic Heart Failure Management. Value Health. 2018 Jul;21(7):772-782. doi: 10.1016/j.jval.2017.11.011. Epub 2018 Mar 21. PMID 30005749
- [Background] Delgoshaei B, Mobinizadeh M, Mojdekar R, Afzal E, Arabloo J, Mohamadi E. Telemedicine: A systematic review of economic evaluations. Med J Islam Repub Iran. 2017 Dec 20;31:113. doi: 10.14196/mjiri.31.113. eCollection 2017. PMID 29951414
- [Background] Kanera IM, Willems RA, Bolman CA, Mesters I, Verboon P, Lechner L. Long-term effects of a web-based cancer aftercare intervention on moderate physical activity and vegetable consumption among early cancer survivors: a randomized controlled trial. Int J Behav Nutr Phys Act. 2017 Feb 10;14(1):19. doi: 10.1186/s12966-017-0474-2. PMID 28187725
- [Background] Galiano-Castillo N, Cantarero-Villanueva I, Fernandez-Lao C, Ariza-Garcia A, Diaz-Rodriguez L, Del-Moral-Avila R, Arroyo-Morales M. Telehealth system: A randomized controlled trial evaluating the impact of an internet-based exercise intervention on quality of life, pain, muscle strength, and fatigue in breast cancer survivors. Cancer. 2016 Oct 15;122(20):3166-3174. doi: 10.1002/cncr.30172. Epub 2016 Jun 22. PMID 27332968
- [Background] Galiano-Castillo N, Arroyo-Morales M, Lozano-Lozano M, Fernandez-Lao C, Martin-Martin L, Del-Moral-Avila R, Cantarero-Villanueva I. Effect of an Internet-based telehealth system on functional capacity and cognition in breast cancer survivors: a secondary analysis of a randomized controlled trial. Support Care Cancer. 2017 Nov;25(11):3551-3559. doi: 10.1007/s00520-017-3782-9. Epub 2017 Jun 22. PMID 28639097
- [Background] Eakin EG, Lawler SP, Winkler EA, Hayes SC. A randomized trial of a telephone-delivered exercise intervention for non-urban dwelling women newly diagnosed with breast cancer: exercise for health. Ann Behav Med. 2012 Apr;43(2):229-38. doi: 10.1007/s12160-011-9324-7. PMID 22109352
- [Background] Demeyer H, Louvaris Z, Frei A, Rabinovich RA, de Jong C, Gimeno-Santos E, Loeckx M, Buttery SC, Rubio N, Van der Molen T, Hopkinson NS, Vogiatzis I, Puhan MA, Garcia-Aymerich J, Polkey MI, Troosters T; Mr Papp PROactive study group and the PROactive consortium. Physical activity is increased by a 12-week semiautomated telecoaching programme in patients with COPD: a multicentre randomised controlled trial. Thorax. 2017 May;72(5):415-423. doi: 10.1136/thoraxjnl-2016-209026. Epub 2017 Jan 30. PMID 28137918
- See also: Treatment stage IV NSCLC (Dutch) — https://www.oncoline.nl/niet-kleincellig-longcarcinoom

DOCUMENTS (1):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03883243/Prot_000.pdf